CLINICAL TRIAL: NCT03303391
Title: Using Intradialytic Systolic Blood Pressure Slopes to Guide Ultrafiltration in Hemodialysis Patients: A Validation Study and Clinical Trial
Brief Title: Using Intradialytic Blood Pressure Slopes to Guide Ultrafiltration
Acronym: IBPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Expired
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Peter Van Buren, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 032017-024
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-03

CONDITIONS: ESRD; Extracellular Fluid Alteration; Hypertension
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): This arm of subjects will have all aspects of fluid management and dialysis management managed by the his/her individual nephrologist
- IBPS Group (Experimental): This group will have ultrafiltration prescriptions dictated by a pre-specified protocol that is based on monthly assessment of intradialytic blood pressure slopes obtained over a two week period.
  Interventions: Other: Intradialytic Blood Pressure Slope Based Ultrafiltration

INTERVENTIONS:
Other: Intradialytic Blood Pressure Slope Based Ultrafiltration — Algorithmic Determination of ultrafiltration based on intradialytic blood pressure slopes calculated at the beginning of each month from the prior two weeks of dialysis treatments
  Arms: IBPS Group

SUMMARY:
This study is an open label randomized clinical trial that comparing intradialytic blood pressure slope-based ultrafiltration prescriptions to standard care in the chronic fluid management of maintenance hemodialysis patients. It also includes a cross sectional component evaluating the associations between intradialytic blood pressure slopes ascertained over 2 week periods with measurements of extracellular water/body weight obtained with multifrequency bioimpedance spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* End Stage Renal Disease on Maintenance Hemodialysis
* Hypertension defined as systolic blood pressure > 140 mmHg pre-dialysis or >130 mmHg post dialysis

Exclusion Criteria:

* Hemodialysis Vintage < 1 month
* Pregnancy
* Nadir Systolic Blood Pressure < 95 mmHg
* Pre or Post dialysis systolic blood pressure > 180 mmHg
* Decrease in systolic blood pressure >60 mmHg from pre to post dialysis
* Ultrafiltration rate >13 mL/kg/hr
* Peridialytic Midodrine Use
* Intradialytic Clonidine use
* Documented Antihypertensive Medication Non-adherence

Bioimpedance will not be peformed on patients with

* amputated arms or legs
* cardiac defibrillator or pacemaker
* presence of metal prostheses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Van Buren, MD, MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Davita Dialysis, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | IBPS Group
Started | 9 | 3
Completed | 9 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to two withdrawals in the intervention group (never began the intervention) the comparison is with 9 vs 3
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | IBPS Group | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 intervention subjects withdrew prior to study intervention starting
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 8 | 2 | 10
    >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to two withdrawals in the intervention group (never began the intervention) the comparison is with 9 vs 3
  years | 53.4 (11) | 57.3 (13) | 54.6 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to two withdrawals in the intervention group (never began the intervention) the comparison is with 9 vs 3
  Participants
    Female | 3 | 2 | 5
    Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to two withdrawals in the intervention group (never began the intervention) the comparison is with 9 vs 3
  Participants
    Hispanic or Latino | 5 | 1 | 6
    Not Hispanic or Latino | 4 | 2 | 6
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to two withdrawals in the intervention group (never began the intervention) the comparison is with 9 vs 3
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 2 | 6
    White | 5 | 1 | 6
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Due to two withdrawals in the intervention group (never began the intervention) the comparison is with 9 vs 3
  Participants
    United States | 9 | 3 | 12
Diabetes [Count of Participants; unit: Participants] — Population: Due to two withdrawals in the intervention group (never began the intervention) the comparison is with 9 vs 3
  Participants | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Ambulatory Systolic Blood Pressure
Description: The change in mean systolic ambulatory blood pressure from study baseline to completion (4 months)
Time Frame: Baseline, 4 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care | IBPS Group
Number analyzed (Participants) | 9 | 3
mmHg | -0.9 (12) | -21.3 (6.7)

2. Secondary Outcome: Change in Extracellular Volume/Body Weight Ratio
Description: expected reduction of at least 0.025 greater reduction for IBPS compared to standard care The change in ECV/body weight from baseline to 4 month
Time Frame: Baseline, 4 months
Population: In the Standard of Care arm/ group, it was not possible to obtain these measurements in 3 subjects (amputations, defibrillators, implanted metal) and are missing the data since they were unable to undergo these measurements.
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Standard Care | IBPS Group
Number analyzed (Participants) | 6 | 3
L/kg | -0.003 (.02) | -.01 (.007)

ADVERSE EVENTS:
Time Frame: Adverse events were determined over a 4 month period per subject
Arm/Group | Standard Care | IBPS Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 5/9 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=9) | IBPS Group (N=3)
Intradialytic Hypotension (Blood and lymphatic system disorders) | 5 (10) | 3 (11) — At least one episode of systolic blood pressure <90 mmHg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03303391/Prot_SAP_000.pdf